CLINICAL TRIAL: NCT03047278
Title: Gabapentin Kinetic Disposition and Renal Excretion: Role of Transporters for Organic Cations and the Effect of Glycemic Control in Patients With Neuropathic Pain.
Brief Title: Transporters for Organic Cations and Glycemic Control in Patients With Neuropathic Pain.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Natalia Valadares de Moraes (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor-Investigator, Natalia Valadares de Moraes, Assistant Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Organization: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBPDIABETCET
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Neuropathic Pain; Type 2 Diabetes Mellitus; Diabetic Neuropathy, Painful
MeSH Terms: conditions — Neuralgia; Diabetes Mellitus, Type 2; Diabetic Neuropathies | interventions — Gabapentin; Cetirizine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Active Comparator): Adult patients (18 - 59 years old) with neuropathic pain of score ≥ 4 that do not use gabapentin were recruited. All patients received oral single dose of gabapentin (300 mg) as capsules after 12 hour-fasting (phase I). To investigate GBP pharmacokinetics, blood samples were collected in heparinized tubes up to 36 hours after GBP administration. The urine of the patients was collected up to 36 hours after GBP administration. The intensity of pain was evaluated in each time of blood sampling through the visual analog scale (0-10). In phase II, after 15 days (wash-out) from phase I, cetirizine hydrochloride (10 mg) was administered orally, twice a day, as pills, for five days. On the last day of cetirizine treatment, an oral single dose of gabapentin (300 mg), as capsule, was administered. Serial blood and urine samples were collected up to 36 hours after GBP administration. The intensity of pain was evaluated in each time of blood sampling.
  Interventions: Procedure: Serial Blood Samples; Procedure: Serial Urine Samples; Drug: Gabapentin 300 mg; Drug: Cetirizine Hydrochloride 10 mg
- Controlled Diabetes Group (Experimental): Adult patients (18 - 59 years old) with controlled type 2 diabetes (glycated hemoglobin ≤ 8.0%) and diabetic neuropathy of score ≥ 4 that do not use gabapentin were recruited. All patients received oral single dose of gabapentin (300 mg) as capsules after 12 hour-fasting. To investigate GBP pharmacokinetics, blood samples were collected in heparinized tubes up to 36 hours after GBP administration. The urine of the patients was collected up to 36 hours after GBP administration. The intensity of pain was evaluated in each time of blood sampling through the visual analog scale (0-10).
  Interventions: Procedure: Serial Blood Samples; Procedure: Serial Urine Samples; Drug: Gabapentin 300 mg
- Uncontrolled Diabetes Group (Experimental): Adult patients (18 - 59 years old) with uncontrolled type 2 diabetes (glycated hemoglobin ≥ 8.0%) and diabetic neuropathy of score ≥ 4 that do not use gabapentin were recruited. All patients received oral single dose of gabapentin (300 mg) as capsules after 12 hour-fasting. To investigate GBP pharmacokinetics, blood samples were collected in heparinized tubes up to 36 hours after GBP administration. The urine of the patients was collected up to 36 hours after GBP administration. The intensity of pain was evaluated in each time of blood sampling through the visual analog scale (0-10).
  Interventions: Procedure: Serial Blood Samples; Procedure: Serial Urine Samples; Drug: Gabapentin 300 mg

INTERVENTIONS:
Procedure: Serial Blood Samples — Serial blood samples were collected at times 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours after gabapentin administration, for all patients.
Procedure: Serial Urine Samples — Serial urine samples were collected at intervals 0-8 hours, 8-16 hours, 16-24 hours and 24-36 hours after gabapentin administration, for all patients.
Drug: Gabapentin 300 mg — All patients were treated with oral single dose of gabapentin 300 mg.
Drug: Cetirizine Hydrochloride 10 mg — Patients of control group were treated with cetirizine hydrochloride, 10 mg, twice as day, orally, for five days.
  Arms: Control Group

SUMMARY:
This study aimed to investigate the influence of the glycemic control of type 2 diabetes (DM2) and of cetirizine (OCTs inhibitor) on gabapentin kinetics disposition and pharmacodynamics (PK-PD) in patients with neuropathic pain. Thus, non-diabetic patients (Control Group, n=10), patients with controlled diabetes (n=9) and patients with uncontrolled diabetes (n=10), all with neuropathic pain of intensity ≥ 4 in pain visual analog scale (0-10) were investigated.

DETAILED DESCRIPTION:
Gabapentin (GBP), anticonvulsant used to neuropathic pain treatment, is mainly eliminated unchanged in urine. Renal active tubular secretion has been suggested to contribute on GBP excretion by renal excretion. Studies performed on rats with experimental diabetes suggest that hyperglycemia reduces the activity of organic cation transporters (Oct). Thus, the aim of the study was to investigate the role of OCTs on kinetic disposition and pharmacodynamics of GBP in patients with neuropathic pain and to verify the regulation of these transporters' activity by glycemic control in diabetes. A cross-over clinical study was performed in patients with neuropathic pain (n=10, Control) to evaluate the influence of CTZ on GBP kinetic disposition. To evaluate the effect of glycemic control, patients with controlled DM2 (DC, n=9) and uncontrolled DM2 (DNC, n=10) were investigated. All participants investigated had neuropathic pain of intensity ≥ 4 evaluated by analogue visual scale (EVA) and were treated with oral single-dose of 300 mg of GBP (Phase 1) or cetirizine (20 mg/day) for 5 days and single-dose of GBP on the last day (Phase 2). Only participants of Control group participated of Phase 2. Serial blood and urine samples were collected up to 36 hours after GBP administration. The intensity of pain was evaluated at the same time of blood sampling, using the visual analog scale. GBP concentration in plasma and urine was validated by JPLC-UV. All participants were genotyped for polymorphisms SLC22A2 808G>T and SLC22A4 1507C>T. The pharmacokinetic parameters were estimated by non-compartmental analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, both gender
* Patients with neuropathic pain with score ≥ 4 in visual analog scale
* Patients with controlled type 2 diabetes (glycated hemoglobin ≤ 8.0%) and diabetic neuropathy with score ≥ 4 in visual analog scale
* Patients with uncontrolled type 2 diabetes (glycated hemoglobin ≥ 8.0%) and diabetic neuropathy with score ≥ 4 in visual analog scale
* Patients that suspend the use of analgesics for 10 times half-life before starting the protocol

Exclusion Criteria:

* Patients with acute or chronicle severe renal failure (creatinine clearance ≤ 30 mL/min)
* Patients with gastrointestinal diseases
* Patients with history of alcohol and drug abuse
* Patients with acute myocardial insufficiency
* Patients with another kind of chronicle pain as severe as neuropathic pain
* Patients in chronicle use of drugs that interact with gabapentin (antacids and cimetidine)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter (AUC) | Up to 36 hours after gabapentin (300 mg) administration
  Area under the plasma concentration versus time (AUC)

SECONDARY OUTCOMES:
Pharmacokinetic parameter (Total clearance) | Up to 36 hours after gabapentin (300 mg) administration
  Total clearance
Pharmacokinetic parameter (Renal clearance) | Up to 36 hours after gabapentin (300 mg) administration
  Renal clearance
Pharmacokinetic parameter (Vd) | Up to 36 hours after gabapentin (300 mg) administration
  Volume of distribution (Vd)
Pharmacokinetic parameter (Elimination half-life) | Up to 36 hours after gabapentin (300 mg) administration
  Elimination half-life

IPD SHARING:
Plan to Share IPD: Undecided